CLINICAL TRIAL: NCT04951297
Title: Development and Validation of a Bowel-routine-based Self Report Questionnaire for Sacral Sparing After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSY201109
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None, just observation — None ,just observation test

SUMMARY:
To develop a self-administered tool for assessment of sacral sparing after spinal cord injury (SCI) and to test its validity in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* patients with SCI

Exclusion Criteria:

* had neurologic impairments unrelated to SCI, such as peripheral nerve injury, brain injury and cognitive deficits, or if they were unable to complete the questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 102
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
sacral sparing self-report questionnaire | 12months
  sacral sparing self-report questionnaire